CLINICAL TRIAL: NCT01098825
Title: Vaccine Hesitancy: A Survey of District VI Pediatric Clinicians
Brief Title: Vaccine Hesitancy: A Survey of Pediatric Clinicians
Status: Completed | Type: Observational
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Christopher Harrison, Children's Mercy Hospitals and Clinics
Other Study IDs: 09 10-218X
Record Dates: First submitted 2010-04-01; First posted 2010-04-05 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Vaccine Hesitancy; Vaccine Refusal
Keywords: vaccine hesitancy; vaccine refusal
MeSH Terms: conditions — Vaccination Hesitancy; Vaccination Refusal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- District VI AAP clinicians
  Interventions: Other: web-based survey

INTERVENTIONS:
Other: web-based survey — Anonymous web-based survey

SUMMARY:
The purpose of this study is to explore the experiences and perceptions of District VI pediatric clinicians on parental vaccine hesitancy and vaccine refusal.

DETAILED DESCRIPTION:
This is a retrospective, convenience sample, descriptive study. Participants will be asked to complete a web-based survey on parental vaccine hesitancy/ vaccine refusal. Survey responses are primarily categorical. Frequencies and averages will be reported using group statistics.

ELIGIBILITY:
Inclusion Criteria:

* Members of District VI American Academy of Pediatrics

Exclusion Criteria:

* Non-English speaking/reading

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: District VI American Academy of Pediatrics clinicians
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2010-04; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J Harrison, MD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States